CLINICAL TRIAL: NCT04274127
Title: Early Screening of Autism Spectrum Disorder in General and Pediatric Practices, Nurseries and Early Child Care Centers, Using Parent Questionnaires and Guidance for Addressing the Child
Brief Title: Early Screening of Autism Spectrum Disorder in General and Pediatric Practices
Acronym: KitCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00823-46
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; screening; ITC; M-CHAT-R
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: estimate the positive predictive value of an early detection kit composed of 2 questionnaires (M-CHAT-R + CSBS-ITC) followed by a confirmation of the detection with a phone call by a neuropsychologist, in children aged 16 to 24 months seen by their usual general practitioner or pediatrician or child care centers or attending nurseries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children aged 16 to 24 (Other): estimate the positive predictive value of an early detection kit composed of 2 questionnaires (M-CHAT-R + CSBS-ITC) followed by a confirmation of the detection with a phone call by a neuropsychologist, in children aged 16 to 24 months seen by their usual general practitioner or pediatrician or child care centers or attending nurseries.
  Interventions: Diagnostic Test: early detection kit composed of 2 questionnaires (M-CHAT-R + CSBS-ITC)

INTERVENTIONS:
Diagnostic Test: early detection kit composed of 2 questionnaires (M-CHAT-R + CSBS-ITC) — completion of 2 questionnaires (M-CHAT-R + CSBS-ITC) followed by a confirmation of the detection with a phone call by a neuropsychologist, in children aged 16 to 24 months seen by their usual general practitioner or pediatrician or child care centers or attending nurseries.
  Other Names: phone call by a neuropsychologist

SUMMARY:
Early screening for Autism Spectrum Disorder has been validated using different screening tools, in particular M-CHAT-R and ITC in different countries. Unfortunaltely, in France, they are not often used. Thus, medium age for diagnosis in France is late. Yet, early interventions has shown efficiency (grade B of HAS 2010 recommendations, HAS 2018) . The American have described an efficient method using partnership between pediatricians and autism specialists (Miller et al). Autism Spectrum Disorders concern 1% of population. The third Autism Plan in France then HAS 2018 Recommandations and The 2018 National Strategy for Autism have propose to implement three levels for early diagnostic : the frontline is constituted by professionals who can detect the firsts signs ( in nurseries, general practice, pediatric practice, early childhood centers), the second line is constituted by the proximity network of professionals who can diagnose " simple " autism ( CMP, CAMSP, neurologic pediatricians), the third line is constituted by expert teem in specialized hospital centers for neurodevelopmental disorders diagnostic.

This organization is, for now, not efficient. First lines professionals are not always formed to autism detection. When the screening is efficient, professionals have difficulties to address children to proximity teem trained to autism diagnostic because of delays or lack of professionals. The second line professionals are note always trained to use diagnostic tools and tend to address all the children to the third line, even when the diagnostic is not complex. The third lign is saturated by all these requests.

DETAILED DESCRIPTION:
The investigator propose to improve autism screening in our region of Rhône-Alpes basing on the detection in nursery, and by first line doctors in order to diagnose autism before 3 year of age. After screening, a specialized teem will realize a follow-up by phone to guide practitioners to a diagnostic teem in proximity. Early screening realized near family house is compulsory to facilitate accessibility and collaboration between professionals. Diagnostic should be realized in a three month delay, conform to the recommendations. Our project proposes to screen the general population of children who hasn't been screened yet for autism.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 16 and 24 months

Exclusion Criteria:

* Patient with previous Autism spectrum disorder (ASD) diagnostic

Ages: 16 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1211 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
number of children with a confirmed ASD diagnosis | V4 (age of 3)
  number of children with a confirmed ASD diagnosis who had an M-CHAT-R and/or CSBS- ITC score confirmed positive at phone call by the neuropsychologist

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Marignier, Principal Investigator — CH Le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No